CLINICAL TRIAL: NCT01955486
Title: Gas Supply, Demand and Middle Ear Gas Balance -- Project 1, Specific Aim 4, Protocol 1
Brief Title: Gas Supply, Demand and Middle Ear Gas Balance -- Preliminary Protocol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Cuneyt M. Alper, Professor, Otolaryngology, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PRO13040671-1; 2P50DC007667 (NIH)
Record Dates: First submitted 2013-09-27; First posted 2013-10-07 (Estimated); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Middle-ear Function
Keywords: flight simulation; middle ear; Eustachian tube function

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- flight simulation (Experimental): flight simulation in pressure chamber
  Interventions: Other: flight simulation

INTERVENTIONS:
Other: flight simulation

SUMMARY:
The purpose of this study is to gather more information on Eustachian tube function and middle-ear pressures during flying. Ten subjects with tympanostomy tubes (plastic tubes inserted in the eardrums) in their ears or holes in their ear-drums will undergo flight simulation in a pressure chamber. Their middle-ear pressures and Eustachian tube function will be monitored at various chamber pressures.

DETAILED DESCRIPTION:
There are individuals who experience severe barotrauma/barotitis during airplane flights and/or free or tanked diving. Previously, one of the investigators modeled the change in middle-ear (ME) pressure during simulated airplane flights for ears with normal Eustachian tube function (ETF) and with different degrees of Eustachian tube (ET) dysfunction (Kanick SC, Doyle WJ. Barotrauma during air travel: predictions of a mathematical model. J Appl Physiol. May 2005;98(5):1592-1602). That model provided a number of important insights into the pathogenesis of ME barotrauma but included two assumptions that have not been validated: 1) in the absence of ET opening, ME pressure is relatively stable (ignoring tympanic membrane volume induced changes) over wide ranges of ambient pressures, and 2) ET periluminal pressures track local ambient pressures. Other, less rigorous, descriptions of ME pressure behavior during flight and diving make different assumptions: 1) ME pressure changes with changes in ambient pressure and 2) ambient and ET mucosa pressures are incompletely coupled. Modeling ME pressure behavior using the two sets of assumptions predicts different ME pressure trajectories and explanations for barotitis/ME barotrauma during flight and diving. Because the behavior of ME pressure during flight (or diving) constrains the interventions that could be used to prevent barotitis/ME barotrauma, it is important to determine which, if either, model is correct.

Ten otherwise healthy subjects aged 18 to 50 years with unilateral or bilateral eardrum perforations or ventilation tubes will be enrolled after obtaining Informed Consent. Complete histories will be taken with a focus on ear-related problems and they will have an ENT examination including tympanometry to document the patency of the ventilation tube and absence of drainage through the tube (disqualifiers). Eligible subjects will be studied in the pressure chamber during a typical flight simulation with periodic interruptions during ascent and descent. During the simulation, one ME will be fitted with an ear-canal probe attached to a pressure transducer and the other with a probe attached to the Forced-Response test system. ME pressure will be continuously monitored in the one ear and the Forced-Response test will be done at chamber pressures of atmospheric, on decreasing pressures (ascent in a flight) at 500 daPa intervals, during stable "cruising" cabin pressure, on increasing pressures (descent in a flight) at 500 daPa intervals and then at atmospheric pressure. All transducers will be referenced to chamber pressure and signals routed via an A-D box to the memory of a computer for on-line display and storage. Outcome variables will consist of the continuous measures of ME pressure in one ear and the periodic measures of ET opening pressure, closing pressure, passive resistance and dilatory efficiency in the contralateral ear.

Under this model, it is expected that, between active/passive ET openings, ME pressure will be relatively stable and not affected by changing chamber pressure and that the measures of ET periluminal pressures (opening pressure, closing pressure and passive resistance) will track chamber pressure.

ELIGIBILITY:
Inclusion Criteria:

* adults 18-50 years of age
* have unilateral or bilateral holes in the eardrums/patent tympanostomy tubes
* otherwise healthy
* ability to read and comprehend English

Exclusion Criteria:

* drainage through either tube or hole in the eardrum
* cold or allergic rhinitis on presentation
* syndrome predisposing to otitis media
* history of ossicular reconstruction

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2018-04-03 (Actual); Study Completion 2018-04-03 (Actual)

PRIMARY OUTCOMES:
middle-ear pressures | single visit
  middle-ear pressure will be monitored continuously during experiment

SECONDARY OUTCOMES:
Eustachian tube function | single visit
  ETF will be measured during simulations

CONTACTS AND LOCATIONS:
Overall Officials: Cuneyt M Alper, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Middle Ear Physiology Laboratory, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No